CLINICAL TRIAL: NCT07194811
Title: Stroke of Unknown Cause: The Impact of Long-term Heart Monitoring on Stroke Recurrence in Women
Brief Title: Stroke of Unknown Cause in Women: The Impact of Long-term Heart Monitoring on Stroke Recurrence
Acronym: STROKEWISE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Haukeland University Hospital (Other); The Dam Foundation (Other); The Norwegian Women´s Public Health Association (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Jannicke Koldaus-Falch, Neurologist and PhD- candidate, University Hospital, Akershus
Other Study IDs: 24/01445
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cryptogenic Stroke; Atrial Fibrillation; Implantable Cardiac Monitor; Secondary Stroke Prevention; Women's Health; Embolic Stroke of Undetermined Source; Oral Anticoagulation
Keywords: Cerebrovascular Disorder; Cardiovascular Disease; Cardiac arrhythmias; Stroke; Ischemic stroke; Atrial Fibrillation; Sex-differences; Women's Health; Secondary Stroke Prevention; Oral anticoagulation; Embolic stroke
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Cerebrovascular Disorders; Cardiovascular Diseases; Arrhythmias, Cardiac; Stroke; Embolic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICM group: Cryptogenic stroke/ESUS with insertable cardiac monitor for detection of atrial fibrillation
- Control group: Non- invasive monitoring and standard of care. Women with cryptogenic stroke(ESUS) from another hospital

SUMMARY:
The goal of this observational study is to investigate sex - differences in detection rate of atrial fibrillation after cryptogenic stroke (embolic stroke of unknown cause) - using an implantable cardiac rhythm monitor - and the treatment effects of oral anticoagulation on recurrent stroke, ischemic cardiovascular events, major bleeding risk, disability and mortality.

The main questions to answer are:

* Is long-term monitoring and detection of atrial fibrillation after stroke of unknown cause in women related to recurrent stroke and disability?
* Is long-term monitoring and initiation of oral anticoagulation related to cardiovascular events and intracranial haemorrhages? And in addition increased in women compared to men?
* Is long-term rhythm monitoring after stroke with unknown cause related to patient reported outcomes in women?

DETAILED DESCRIPTION:
This is a prospective, observational, study including consecutive patiens with acute cryptogenic stroke /embolic stroke of unknown source (ESUS) or transient ischemic attack (TIA) admitted between 2016 and 2023 at Akershus University Hospital (AUH). As part of the standard investigation at AUH, selected patients are offered an implantable cardiac monitor (ICM) and followed up for detection of atrial fibrillation (AF) by a specialised neurocardiology team. A control group recruited at another hospital during the same period, Haukeland University Hospital (HUS), only comprise women.

The primary objectives:

* To investigate among women with stroke of unknown cause, the effect of implantable cardiac monitors compared to standard non-invasive approach on AF detection, recurrent stroke, death and disability.
* To investigate sex- differences in patients with stroke of unknown cause, the effect of implantable cardiac monitors on AF detection, recurrent stroke, death and disability.

Secondary objectives:

* To compare the rate of cardiovascular events and intracranial haemorrhages after stroke of unknown cause in women offered implantable cardiac monitors, compared to best standard non-invasive follow up
* To investigate the impact of implantable cardiac monitors on the use of oral anticoagulation in women
* To investigate self-perceived health and health related quality of life after stroke of unknown cause in women offered implantable loop recorders, compared to women offered best standard non-invasive approach to detect AF

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cryptogenic stroke or TIA, according to the TOAST (Trial of Org 10172 in Acute Stroke Treatment) classification and an implantable cardiac rythm monitor (ICM) for the ICM group not the control

Exclusion Criteria:

* Patients with known or newly detected AF on standard ECG or 24 h Holter ECG.
* Patients on oral anticoagulants (OAC) for non-AF indications
* Patients with strong contraindications for OAC
* Severe cognitive impairment or disability or with a short life expectancy due to comorbidities of less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total 1050 patients. A cohort of at least 700 patients of both sexes diagnosed with acute cryptogenic stroke or TIA and with an implantable cardiac monitor, admitted to the stroke unit at Akershus University Hospital, Norway.
  A control group of 350 women with acute cryptogenic stroke or TIA, with non-invasive standard monitoring, admitted to the stroke unit at Haukeland University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation deteceted after stroke and transient ischemic attack (TIA) | 30 days and 1 year after index stroke
  >30 seconds of atrial fibrillation detection using implantable cardiac monitor/implantable loop-recorder
Recurrent ischemic stroke after 1 and 2 years | 30 days, 1 and 2 years after index stroke
  Ischemic stroke/TIA: Clinical diagnosis (TOAST criteria) verified by CT and/or MR.

SECONDARY OUTCOMES:
Composite of stroke and mortality | 30 days, 1 and 2 years after index stroke
  Ischemic and heamorragic stroke, (ICD-10 I63 and I61) transient ischemic attack(TIA) (ICD10: G45.9) and mortality
Intracranial bleeding | 30 days, 1 and 2 years after index stroke
  Symptomatic intracranial heamorrage (stroke) (ICD-10: I61)
Patient Reported Outcome Measureres | 3 months after index stroke
  Self-perceived health and health related quality of life by using the EuroQol scale (EQ-5D-5L)
Ischemic cardiac events | 1 and 2 years
  Hospitaized for ischemic cardiac events (ICD10 20-25)
Safety outcome | 1 and 2 years after index stroke
  Hospitalized for gastrointestinal bleeding (ICD 10 K92) and/or intracranial bleeding (I61)
Oral anticoagulation | 1 and 2 years
  Use of oral anticoagulation
Functional outcome 3 months post-stroke | 3 months after index stroke
  Functional outcome 3 months post-stroke using modified Rankin Scale (mRS) from the national stroke registry

CONTACTS AND LOCATIONS:
Overall Officials: Ole Morten Rønning, Professor, Study Director — Akerhus University Hospital and University of Oslo
Locations (1):
- Akershus University Hospital, Department of Neurology, Oslo, Lørenskog/Akershus, Norway

IPD SHARING:
Plan to Share IPD: No
Due to Norwegian regulations, the data cannot be shared publicly, and the authors are not permitted to share the data or study materials used in this study. De-identified datasets may be made available from the corresponding author upon reasonable request and with appropriate ethical and institutional approvals.

REFERENCES:
- [Background] Skrebelyte-Strom L, Ronning OM, Dahl FA, Steine K, Kjekshus H. Prediction of occult atrial fibrillation in patients after cryptogenic stroke and transient ischaemic attack: PROACTIA. Europace. 2022 Dec 9;24(12):1881-1888. doi: 10.1093/europace/euac092. PMID 35819199